CLINICAL TRIAL: NCT03007732
Title: Phase 2 Trial Pembrolizumab or Pembrolizumab in Combination With Intratumoral SD-101 Therapy in Patients With Hormone-Naïve Oligometastatic Prostate Cancer Receiving Stereotactic Body Radiation Therapy and Intermittent Androgen Deprivation Therapy
Brief Title: Pembrolizumab +/- SD-101 in Hormone-Naïve Oligometastatic Prostate Cancer With RT and iADT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Oh (Other)
Collaborators: Prostate Cancer Foundation (Other); Merck Sharp & Dohme LLC (Industry); TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David Oh, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16703; NCI-2017-01340 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2016-08-05; First posted 2017-01-02 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab; Toll-Like Receptor 9; Leuprolide; Abiraterone Acetate; Prednisone; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) (Experimental): Three month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + abiraterone by mouth daily with prednisone by mouth daily (or equivalent medication per local standard practice) for 9 months starting on Day 1.
  Pembrolizumab: Given IV every 21 days for up to 13 doses
  Radiotherapy: Given every other day over 10-14 days delivered to the whole prostate gland via stereotactic body radiation therapy (SBRT) starting 1-2 weeks after marker placement.
- Cohort 1, Arm 2: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) (Experimental): Three month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + abiraterone by mouth daily with prednisone by mouth daily (or equivalent medication per local standard practice) for 9 months starting on Day 1.
  TLR9 agonist SD-101: Injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1
  Pembrolizumab: Given IV every 21 days for up to 13 doses
  Radiotherapy: Given every other day over 10-14 days delivered to the whole prostate gland via stereotactic body radiation therapy (SBRT) starting 1-2 weeks after marker placement.
- Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) (Experimental): Three month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + abiraterone by mouth daily with prednisone by mouth daily (or equivalent medication per local standard practice) for 9 months starting on Day 1.
  Pembrolizumab: Given IV every 21 days for up to 13 doses
  Radiotherapy: Given every other day over 10-14 days delivered to the whole prostate gland and oligometastatic sites via stereotactic body radiation therapy (SBRT) starting 1-2 weeks after marker placement.
  Interventions: Drug: Pembrolizumab; Drug: Leuprolide acetate; Drug: Abiraterone Acetate; Drug: Prednisone; Radiation: Stereotactic Body Radiation Therapy
- Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101) (Experimental): Three month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + abiraterone by mouth daily with prednisone by mouth daily (or equivalent medication per local standard practice) for 9 months starting on Day 1.
  TLR9 agonist SD-101: Injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1
  Pembrolizumab: Given IV every 21 days for up to 13 doses
  Radiotherapy: Given every other day over 10-14 days delivered to the whole prostate gland and oligometastatic sites via stereotactic body radiation therapy (SBRT) starting 1-2 weeks after marker placement.
  Interventions: Drug: Pembrolizumab; Drug: SD-101; Drug: Leuprolide acetate; Drug: Abiraterone Acetate; Drug: Prednisone; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV every 21 days for up to 13 doses (Arms 1 and 2)
  Other Names: MK-3475; Keytruda
  Arms: Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Drug: SD-101 — 5 mg will be delivered to the dominant prostatic tumor lesion at time of fiducial marker placement (1-5 weeks prior to Cycle 1, Day 1) and and 1-3 weeks after Cycle 1 Day 1
  Other Names: Toll-like receptor 9
  Arms: Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Drug: Leuprolide acetate — 22.5 mg will be given intramuscularly (IM). First injection 3 months prior to Cycle 1 Day 1. Intermittent androgen deprivation therapy will be given every 3 months starting Cycle 1, Day 1 for 3 additional doses.
  Other Names: Intermittent androgen deprivation therapy
  Arms: Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Drug: Abiraterone Acetate — 1000 mg oral dosage will be given daily for 3 months prior to Cycle 1, Day 1 and daily for 9 months starting Cycle 1, Day 1.
  Other Names: Intermittent androgen deprivation therapy
  Arms: Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Drug: Prednisone — 5 mg oral dosage will be given daily for 3 months prior to Cycle 1 Day 1 and daily for 9 months starting Cycle 1, Day 1.
  Other Names: Intermittent androgen deprivation therapy
  Arms: Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Radiation: Stereotactic Body Radiation Therapy — 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days.
  Other Names: SBRT
  Arms: Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)

SUMMARY:
This is a non-comparative open-label multicenter Phase 2 clinical trial combining stereotactic body radiation therapy (SBRT) and pembrolizumab with or without intratumoral SD-101 in participants with newly diagnosed hormone-naive oligometastatic prostate cancer.

DETAILED DESCRIPTION:
This randomized phase II trial studies how well androgen deprivation therapy, pembrolizumab, and stereotactic body radiation therapy with or without toll-like receptor 9 (TLR9) agonist SD-101 in treating participants with prostate cancer and cancer in all oligometastatic sites that has spread to other places in the body. Androgen can cause the growth of tumor cells. Androgen deprivation therapy, such as leuprolide acetate, prednisone, and abiraterone acetate may lessen the amount of androgen made by the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Colony-stimulating factors, such as TLR9 agonist SD-101, may increase the production of blood cells. It is not yet known whether giving androgen deprivation therapy, pembrolizumab, and stereotactic body radiation therapy with or without TLR9 agonist SD-101 may work better in treating participants with prostate cancer and cancer in all oligometastatic sites.

PRIMARY OBJECTIVES

COHORT 1:

-- To assess the safety associated with giving RT and pembrolizumab with or without intratumoral SD-101.

COHORT 2:

* To continue to assess the safety associated with giving RT and pembrolizumab with or without intratumoral SD-101.
* To assess if the rate of PSA < nadir + 2 ng/mL at 15 months in participants with non-castrate levels of testosterone is greater than the historical control in each study arm.

SECONDARY OBJECTIVES

COHORT 2 ONLY:

* To determine the rate of testosterone-prostate specific antigen (PSA) uncoupling in each study arm in Cohort 2. Testosterone-PSA uncoupling is defined as PSA < 50% baseline and < 20ng/mL for at least 3 months after testosterone recovers to >150 ng/dL. In participants with metastatic hormone sensitive prostate cancer off hormonal therapy, >90% of participants are expected to have PSA increase to > 50% baseline after 3 months of testosterone recovery.
* To estimate time to clinical progression in each study arm in Cohort 2.
* To estimate progression-free survival (PFS) in each study arm Cohort 2.

EXPLORATORY OBJECTIVE

* To assess peripheral and tumor-based biomarkers of response and resistance in both cohorts.
* To define the treatment-induced effects on circulating immune cells in both cohorts.
* To explore remodeling of circulating T cell repertoire in both cohorts.
* To explore the concordance of Prostate-Specific Membrane Antigen (PSMA) - Positron Emission Tomography (PET) scanning with conventional imaging in oligometastatic prostate cancer participants in both cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >=18 years of age on day of signing informed consent.
3. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
4. Histologically documented adenocarcinoma of the prostate
5. Oligometastatic disease. In order to be eligible, the participant must have a total of <4 metastatic bone and/or metastatic lymph node sites based on bone and/or soft tissue lesions as defined by any of the following:

   1. Bone metastases will be defined by bone imaging. If the participant has technetium bone scan, and/or sodium fluoride (NaF) PET performed, either study may be used for documenting metastases; both scans do not need to show the number of metastases required for study entry. For participants undergoing PSMA PET, only PSMA avid lesions that are consistent with metastasis will be counted as a site of metastasis.
   2. Distant metastatic lymph node disease. A lymph node ≥1 cm in shortest dimension will be noted as involved with disease. Distant metastatic lymph nodes will be determined as any lymph nodes outside the confines of the true pelvis. For participants undergoing PSMA PET, only PSMA avid lesions that are consistent with metastasis will be counted as a site of metastasis.
   3. Any other soft tissue lesion deemed by the physician to be consistent with distant metastatic disease. For participants undergoing PSMA PET, only PSMA avid lesions that have a CT or MRI correlate consistent with metastasis will be counted as a site of metastasis.

      * Note: Radiographic imaging performed as standard of care prior to obtaining informed consent and within 60 days of initiating study treatment may be used to assess oligometastatic disease during screening, rather than repeating scans. For participants who have started on ADT, they must have had imaging prior to initiation of hormonal therapy
6. Treatment naïve, defined as less than 2 months of standard of care ADT (e.g. GnRH agonist or antagonist with or without antiandrogen, including abiraterone) for metastatic hormone-sensitive prostate cancer prior to enrollment (at the time of consent)
7. No prior chemotherapy for prostate cancer
8. Not a candidate for or refuse chemotherapy
9. No prior prostatectomy or prostatic radiation
10. PSA >2 ng/mL at baseline or prior to initiation of hormonal therapy
11. Baseline testosterone >150 ng/dL if participant has not initiated hormonal therapy, for those participants who have already initiated hormonal therapy, baseline testosterone is not required
12. Consent to undergo mandatory prostatic core biopsies at the time of fiducial marker placement and 1-3 weeks after Cycle 1 Day 1 of pembrolizumab.
13. The effects of pembrolizumab on the developing human fetus is unknown. Men treated or enrolled on this protocol must agree to use adequate contraception prior to the first dose of study therapy, for the duration of the study participation, and for 120 days after the last dose of study therapy. Their partners should also be encouraged to use proper method of contraception. Their partners should also be encouraged to use proper method of contraception.
14. Demonstrate adequate organ function defined as: Adequate Organ Function Laboratory Values (Performed within 10 days of treatment initiation):

    * Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL)
    * Platelets >=100,000 / mcL
    * Hemoglobin >=9 g/dL or ≥5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
    * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) <=1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. Creatinine clearance should be calculated per institutional standard
    * Serum total bilirubin <= 1.5 X ULN OR Direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 ULN
    * Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
    * Albumin >2.5 mg/dL
    * International Normalized Ratio (INR) or Prothrombin Time (PT)
    * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

1. Participants who are not appropriate candidates for prostate or oligometastasis-directed SBRT
2. Participants with neuroendocrine or small cell features are not eligible.
3. Participants with evidence of liver metastasis are excluded.
4. Gonadotropin-releasing hormone (GnRH) agonists or GnRH antagonists (e.g., leuprorelin, degarelix) for > 2 months prior to consenting
5. Antiandrogens (e.g., bicalutamide, flutamide, nilutamide, abiraterone, enzalutamide) for > 2 months prior to consenting. Participants on 5-alpha reductase inhibitors are allowed on study.
6. Estrogen containing compounds for > 2 months prior to consenting
7. PC-SPES or PC-x products. Other herbal therapies or supplements will be considered by the Principle Investigator on a case-by-case basis based on their potential for hormonal or anti-cancer therapies.
8. Prior immunotherapy or chemotherapy for prostate cancer
9. Prior radiation therapy to the prostate
10. Prior prostatectomy
11. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
12. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment, with the exception of steroids for adrenal insufficiency in which case prednisone =<10mg/day or its equivalent is allowed.
13. Has a known history of active Bacillus Tuberculosis (TB)
14. Hypersensitivity to pembrolizumab or any of its excipients.
15. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
16. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

    * Note: Subjects with <= Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
    * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting
17. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include carcinoid, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
18. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroid treatment for at least 14 days prior to the first dose of study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
19. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
20. Has known history of, or any evidence of active, non-infectious pneumonitis.
21. Has an active infection requiring systemic therapy.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
24. Expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
25. Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1) , or anti-Programmed cell death 1 ligand 2 (PD-L2) agent.
26. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
27. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV) (i.e. HCV RNA [qualitative] is detected).
28. Has received a live vaccine within 30 days of planned start of study therapy. a. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Oh, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab); Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab): Three-month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + 1000 mg oral daily with 5mg oral prednisone daily (or equivalent medication per local standard practice) for 9 months starting on Day 1. Pembrolizumab: 200 mg IV every 21 days for up to 13 doses, stereotactic body radiation therapy (SBRT) 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days.
- Cohort 1, Arm 2: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101): Three-month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + 1000 mg oral daily with 5mg oral prednisone daily (or equivalent medication per local standard practice) for 9 months starting on Day 1. Pembrolizumab: 200 mg IV every 21 days for up to 13 doses, stereotactic body radiation therapy (SBRT) 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days. TLR9 agonist SD-101 will be injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1.
- Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101): Three-month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + 1000 mg oral daily with 5mg oral prednisone daily (or equivalent medication per local standard practice) for 9 months starting on Day 1. Pembrolizumab: 200 mg IV every 21 days for up to 13 doses, stereotactic body radiation therapy (SBRT) 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days. Toll-like receptor 9 (TLR9) agonist SD-101 will be injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) | Cohort 1, Arm 2: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Started | 5 | 5 | 7 | 6
Completed | 5 | 5 | 6 | 5
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal from study post randomization but just prior to receiving any treatment | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two participants in Cohort 2 withdrew from the study immediately after randomization and prior to receiving any study treatment. Having not received any investigational treatment, the two participants were not evaluable for analysis per protocol, and have been removed from the baseline analysis population.
Groups:
- Cohort 2, Arm 2: Prostate and Oligometastatic Sites (ADT, SBRT, Pembrolizumab, SD-101): Three-month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + 1000 mg oral daily with 5mg oral prednisone daily (or equivalent medication per local standard practice) for 9 months starting on Day 1. Pembrolizumab: 200 mg IV every 21 days for up to 13 doses, stereotactic body radiation therapy (SBRT) 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days. TLR9 agonist SD-101 will be injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) | Cohort 1, Arm 2: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) | Cohort 2, Arm 1: Prostate and Oligometastatic Sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic Sites (ADT, SBRT, Pembrolizumab, SD-101) | Total
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 21
Age, Continuous [Mean (Full Range); unit: years old] | 67 [61 to 72] | 63 [53 to 73] | 66.8 [59 to 70] | 72.2 [57 to 83] | 67.2 [53 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 6 | 5 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 6 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 6 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change Rate of Prostate-specific Antigen (PSA) < Nadir + 2 ng/mL From First Day of Treatment to 15 Months (Cohort 2)
Description: Only participants in cohort 2, who achieve testosterone recovery to non-castrate levels (>150 ng/dL) at 15 months, will be analyzed for the primary endpoint. The rate of PSA < nadir + 2 ng/mL at 15 months from the start of radiotherapy and cycle 1, day 1 of pembrolizumab, among participants whose testosterone recovers to non-castrate levels (>150 ng/dL). The point estimate of the rate of PSA < nadir + 2 ng/mL will be obtained with its 95% confidence interval for participants by arm in cohort 2. All participants who receive any part of a dose of RT, SD-101 or pembrolizumab will be analyzed for efficacy.
Time Frame: Start of treatment and 15 months (approx. 15 months total)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Number analyzed (Participants) | 6 | 5
percentage of participants | 100 [54.1 to 100] | 100 [47.8 to 100]

2. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Adverse events occurring on study will be summarized for all participants that received study intervention (including pembrolizumab, SD-101, SBRT to prostate, SBRT to oligometastatic sites) by maximum toxicity grade across study arms.
Time Frame: Up to 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) | Cohort 1, Arm 2: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Number analyzed (Participants) | 5 | 5 | 6 | 5
Participants
  Acute kidney injury, Grade 2 | 1 | 0 | 0 | 0
  Adrenal Insufficiency, Grade 2 | 1 | 0 | 0 | 0
  Alanine aminotransferase increased, Grade 3 | 2 | 1 | 0 | 1
  Alkaline phosphatase increased, Grade 2 | 0 | 0 | 0 | 1
  Anemia, Grade 1 | 0 | 2 | 1 | 0
  Arthralgia, Grade 2 | 0 | 0 | 0 | 1
  Arthritis, Grade 2 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased, Grade 3 | 2 | 1 | 0 | 1
  Blood bilirubin increased, Grade 2 | 1 | 1 | 0 | 0
  Chills, Grade 1 | 0 | 2 | 0 | 0
  Colitis, Grade 3 | 1 | 1 | 0 | 1
  Creatinine increased, Grade 2 | 1 | 0 | 0 | 0
  Cystitis noninfective, Grade 2 | 0 | 0 | 1 | 0
  Depression, Grade 1 | 0 | 0 | 0 | 1
  Diarrhea, Grade 3 | 0 | 0 | 0 | 1
  Dry mouth, Grade 1 | 1 | 0 | 0 | 0
  Dysphagia, Grade 1 | 0 | 0 | 0 | 1
  Fatigue, Grade 2 | 0 | 0 | 1 | 0
  Fever, Grade 1 | 0 | 2 | 0 | 0
  Flu-like symptoms, Grade 1 | 0 | 1 | 0 | 0
  Gynecomastia, Grade 2 | 0 | 0 | 1 | 0
  Headache, Grade 1 | 0 | 1 | 0 | 2
  Hematuria, Grade 2 | 0 | 0 | 1 | 0
  Hot flashes, Grade 1 | 0 | 0 | 0 | 1
  Hyperglycemia, Grade 1 | 0 | 0 | 1 | 0
  Hypertension, Grade 2 | 0 | 0 | 1 | 1
  Hypokalemia, Grade 3 | 0 | 0 | 1 | 0
  Hypothyroidism, Grade 2 | 0 | 0 | 1 | 0
  Infusion related reaction, Grade 1 | 0 | 1 | 0 | 0
  Localized edema, Grade 1 | 1 | 0 | 0 | 0
  Mucositis oral, Grade 1 | 0 | 2 | 1 | 0
  Musculoskeletal and connective tissue disorder - Other, specify | 0 | 0 | 0 | 1
  Myalgia, Grade 1 | 0 | 3 | 0 | 1
  Nausea, Grade 2 | 0 | 0 | 0 | 1
  Platelet count decreased, Grade 1 | 0 | 0 | 1 | 0
  Proctitis, Grade 2 | 0 | 0 | 1 | 2
  Pruritus, Grade 1 | 0 | 0 | 1 | 0
  Rash maculo-papular, Grade 3 | 0 | 3 | 0 | 0
  Rectal hemorrhage, Grade 1 | 0 | 1 | 0 | 0
  Renal and urinary disorders - Other, specify, Grade 1 | 0 | 0 | 1 | 0
  Sneezing, Grade 1 | 0 | 0 | 0 | 1
  Urinary frequency, Grade 1 | 1 | 0 | 0 | 0
  Urinary retention, Grade 1 | 0 | 0 | 0 | 2
  Urticaria, Grade 1 | 0 | 0 | 0 | 1
  Vomiting, Grade 2 | 0 | 0 | 1 | 0
  Weight Gain, Grade 1 | 0 | 0 | 0 | 1

3. Secondary Outcome: Rate of Testosterone-PSA Uncoupling (Cohort 2)
Description: Testosterone-PSA uncoupling is defined as PSA < 50% baseline and < 20ng/mL for at least 3 months after testosterone recovers to >150 ng/dL. In participants with metastatic hormone-sensitive prostate cancer off hormonal therapy, >90% participants are expected to have PSA increase to > 50% baseline after 3 months of testosterone recovery. Therefore, the presence of PSA testosterone uncoupling in this study may serve as a surrogate of immunotherapeutic responses induced by pembrolizumab combined with RT (arm 1), or RT with SD-101 (arm 2), if a prolonged PSA < nadir + 2 ng/mL is not achieved. The point estimate of testosterone-PSA uncoupling rate will be obtained with its 95% confidence interval for each arm in cohort 2.
Time Frame: Up to 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Number analyzed (Participants) | 6 | 5
percentage of participants | 66.7 [22.3 to 95.7] | 80 [28.4 to 99.5]

4. Secondary Outcome: Median Time to Clinical Progression (Cohort 2)
Description: The time to clinical progression in each study arm in cohort 2 is defined as the time to radiographic progression by Prostate Specific Antigen Working Group-2 (PSAWG2) criteria, time to symptomatic progressive disease, or PSA progression, whichever comes the first. Kaplan-Meier estimate will be obtained for the time to clinical progression in each study arm in cohort 2
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Number analyzed (Participants) | 6 | 5
months | NA [23.5 to NA] — There was an insufficient number of events therefore a median and upper limit could not be calculated | 25.4 [19.8 to NA] — There was an insufficient number of events therefore an upper limit could not be calculated

5. Secondary Outcome: Median Progression-free Survival (PFS) (Cohort 2)
Description: Progression-free survival (PFS) will be estimated for each study arm on cohort 2 by Kaplan-Meier estimate, where PFS is a composite endpoint based on PSA progression, radiological progression, clinical deterioration, or death.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
Number analyzed (Participants) | 6 | 5
months | NA [23.5 to NA] — There was an insufficient number of events therefore a median and upper limit could not be calculated | 25.4 [19.8 to NA] — There was an insufficient number of events therefore an upper limit could not be calculated

ADVERSE EVENTS:
Time Frame: Up to 3 years
Groups:
- Cohort 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101); Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101): Three-month androgen deprivation therapy (ADT) run-in followed by leuprolide injected intramuscularly every 3 months for 3 doses (or another FDA approved gonadotropin-releasing hormone agent for 9 months) + 1000 mg oral daily with 5mg oral prednisone daily (or equivalent medication per local standard practice) for 9 months starting on Day 1. Pembrolizumab: 200 mg IV every 21 days for up to 13 doses, stereotactic body radiation therapy (SBRT) 7 Gy x 5 fractions (35 Gy total) 1-2 weeks after fiducial marker placement and simulation over 10-14 days. TLR9 agonist SD-101 will be injected into the dominant prostatic tumor lesion at time of fiducial marker placement (1-5weeks prior to Cycle 1 Day 1) and 1-3 weeks after Cycle 1 Day 1.
Arm/Group | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) | Cohort 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/6 | 1/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) (N=5) | Cohort 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) (N=5) | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) (N=6) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101) (N=5)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab) (N=5) | Cohort 1: Prostate Only Sites (ADT, SBRT, Pembrolizumab, SD-101) (N=5) | Cohort 2, Arm 1: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab) (N=6) | Cohort 2, Arm 2: Prostate and Oligometastatic sites (ADT, SBRT, Pembrolizumab, SD-101) (N=5)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (6) | 1 (1) | 0 (0) | 1 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (5) | 2 (3) | 3 (4) | 5 (5)
Pain (General disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatobilliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications, Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (8) | 2 (3) | 2 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 3 (9) | 1 (2) | 0 (0) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (3) | 2 (2) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Weight Gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 2 (3) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized edema (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (5) | 2 (2) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 0 (0) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (8) | 2 (2)
Hot Flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03007732/Prot_SAP_000.pdf